CLINICAL TRIAL: NCT07094230
Title: Combination iSTAT/Alinity and IR Oculography for Head CT Necessity and Recovery Prediction After mTBI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Captain James A. Lovell Federal Health Care Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jim Buskirk PT, DPT, PhD, MS Ed, Co-Investigator, Captain James A. Lovell Federal Health Care Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1850604
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Blood
Keywords: mTBI; biomarkers; IR Oculography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- blood biomarkers analyses (Experimental): blood biomarkers analyses
  Interventions: Diagnostic Test: biomarkers analyses

INTERVENTIONS:
Diagnostic Test: biomarkers analyses — blood analyses

SUMMARY:
Use of blood biomarkers and eye tracking after traumatic brain injury for recovery timeline prediction

DETAILED DESCRIPTION:
Use of blood biomarkers and video IR oculography after mTBI for necessity of head CT scan and recovery timeline prediction

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-85, Communicative in English language, With clinician-confirmed mTBI (GCS 13-15, ≤24 hours post-injury)

Exclusion Criteria:

Neurological, vestibular, or visual disorders, Significant comorbidities, Prior TBI (<6 months) Special populations (pregnant, incarcerated, active-duty recruits). Active-duty recruits excluded due to inability to contact them at scheduled intervals for remote follow-up questionnaires.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
blood biomarkers analyses | same day
  Alinity device analyses of GFAP and UCH-L1

CONTACTS AND LOCATIONS:
Overall Officials: James Buskirk, PT, DPT, PhD, MS, Study Director — Captain James A. Lovell Federal Health Care Center
Locations (1):
- Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
blood analyses results, IR Oculography results, recovery timelines questionnaires data
Supporting Information: SAP
Time Frame: August 1, 2025 -- August 1, 2026
Access Criteria: Rosalind Franklin University Dept of Statistics, IPD, via electronic data transfer
URL: https://department.va.gov/administrations-and-offices/enterprise-integration/data-governance-and-analytics/

REFERENCES:
- See also: Blood biomarkers analyses — https://www.corelaboratory.abbott/int/en/offerings/brands/alinity.html